CLINICAL TRIAL: NCT01496586
Title: Fatigue and Amotivation Following Mild Traumatic Brain Injury and Their Influence on Service Member Community Reintegration
Brief Title: Service Member Fatigue and Lack of Motivation Following Concussion
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120030; 12-N-0030
Record Dates: First submitted 2011-12-17; First posted 2011-12-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-08-03

CONDITIONS: Fatigue; Traumatic Brain Injury
Keywords: Fatigue; Traumatic Brain Injury; Motivational Incentive; TBI
MeSH Terms: conditions — Fatigue; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Many service members have reported feeling tired, a loss of motivation, mood changes, and problems working with others after they have a concussion during deployment. These problems may lead to problems with their job and relationships. This study hopes to figure out what parts of the brain may be affected in people with these problems after a concussion.

Objectives:

- To learn more about the problems that may occur after service members have a concussion during deployment and return home.

Eligibility:

* Service members or veterans between 18 and 40 years of age who have had a mild traumatic brain injury (concussion) in the past 6 months.
* Companions (at least 18 years of age) of the service members will also be included in this study. Companions will have interacted with the service member at least 1 hour a week since deployment.

Design:

* Service members will have 1 week of tests at the National Institutes of Health Clinical Center. Companions will have 2 days of tests at the Center.
* Each day, service members will have 4 or 8 hours of tests. Tests will include a medical history and physical exam, neuropsychological tests and imaging studies. The tests will ask about fatigue, stress, mood, pain, daily activities, and family support. The imaging studies will measure brain function at rest and during activity.
* Companions will have a medical history and physical exam. They will also complete several questionnaires about themselves as well as the service member/veteran. The tests will ask about fatigue, stress, mood, pain, daily activities, and family support....

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to determine the behavioral-anatomical relationships that underlie fatigue and amotivation following mild traumatic brain injury in deployed military service members. The specific aims are to 1) determine the neural correlates of fatigue, and 2) assess how fatigue and social cognition relate to social outcomes including employment, community integration and participation in social activities. The theory we will test is that fatigue in this population is the result of subtle changes in frontal cortical and subcortical structures.

Study Design: Observational, natural history study.

Populations: 1) Individuals who have sustained a mild traumatic brain injury as a service member deployed in support of Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn, and who continue to experience symptoms more than 6 months after injury, and 2) Companions of individuals from the first group.

Outcome Measures: We will seek statistical associations between fatigue measures and brain morphometric and white matter diffusion measurements obtained by MRI as well as task and resting state fMRI.

ELIGIBILITY:
* INCLUSION CRITERIA mTBI GROUP:
* Diagnosis of at least one mTBI during deployment;
* At least six months from time of injury;
* Age range 18 or older;
* A self-report of somatic or behavioral symptoms that developed within 3 months following mTBI and were not present before injury, and may or may not be present at enrollment:

  * Easy fatiguability
  * Sleep disturbance
  * Headache or other chronic widespread pain that does not seem related to extremity injury
  * Emotional lability
  * Lack of spontaneity or apathy
  * Lack of motivation
  * Feelings of anxiety
  * Personality change that they or others have noticed
  * Irritability or aggressiveness
* The mTBI participant provides informed consent.

EXCLUSION CRITERIA mTBI GROUP:

* Daily use of stimulants, narcotics, hypnotic or anxiolytics
* Diagnosis of sleep apnea, thyroid disorder, or rheumatoid arthritis
* Any history of head injury associated with a loss of consciousness that lasted longer than 24 hours (not including sedation);
* Daily use of more than 600mg caffeine (equivalent to approximately five cups of coffee).
* Headaches more than once a month prior to deployment;
* Pregnancy;
* Claustrophia;
* Inability to comfortably lie supine for two hours

INCLUSION CRITERIA companion group

* Chosen by a mTBI participant as a close companion (i.e, spends or in the last 3 years has spent a minimum of 1 hour per week on average with the mTBI participant and with whom the mTBI participant is comfortable discussing personal matters);
* The companion provides informed consent.

EXCLUSION CRITERIA companion group:

-Lack of understanding of the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-12-01; Study Completion 2015-08-03

PRIMARY OUTCOMES:
Correlations between fractional anisotropy, effective connectivity measured by size of cortical and subcortical structures on DTI, and VBM that correlate with measures of fatigue, apathy, effort expenditure. | One year

SECONDARY OUTCOMES:
Correlations between fractional anisotropy, effective connectivity measured by size of cortical and subcortical structures on DTI, and VBM that correlate with measures of alexithymia and perceived stress | One year

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750
- [Background] Jones E, Fear NT, Wessely S. Shell shock and mild traumatic brain injury: a historical review. Am J Psychiatry. 2007 Nov;164(11):1641-5. doi: 10.1176/appi.ajp.2007.07071180. PMID 17974926
- [Background] Jones E, Hodgins-Vermaas R, McCartney H, Everitt B, Beech C, Poynter D, Palmer I, Hyams K, Wessely S. Post-combat syndromes from the Boer war to the Gulf war: a cluster analysis of their nature and attribution. BMJ. 2002 Feb 9;324(7333):321-4. doi: 10.1136/bmj.324.7333.321. PMID 11834557